CLINICAL TRIAL: NCT02867670
Title: TMS as a Biological Marker of Neuroplasticity
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 818784
Record Dates: First submitted 2016-06-03; First posted 2016-08-16 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Stroke; Aphasia
Keywords: Transcranial Magnetic Stimulation (TMS)
MeSH Terms: conditions — Stroke; Aphasia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The investigators are asking participants to provide a saliva sample which will later be genotyped for the BDNF protein.
  Saliva samples are optional.

GROUPS / COHORTS (2):
- Transcranial Magnetic Stimulation of Motor Cortex: All study participants will receive real TMS stimulation over the primary motor cortex in order to collect physiological measures which will later be correlated with measures of neuroplasticity. There is NO placebo stimulation.
  Interventions: Device: Transcranial Magnetic Stimulation
- Transcranial Magnetic Stimulation of Language Cortex: All study participants will receive real TMS stimulation over the language cortex and a control site (i.e. vertex). Transient changes in speech production will be recorded and compared to measures of neuroplasticity. There is NO placebo stimulation.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — TMS is a form of non-invasive brain stimulation which uses magnetic pulses to stimulate regions of the brain from outside the head, on the scalp. Specifically, TMS is performed with a copper-and-plastic coil that emits a magnetic field, which can affect brain cells in specific locations. In this study, researchers will also use a form of TMS called theta-burst stimulation (TBS), where TMS pulses are delivered rapidly over time.
  Other Names: TMS

SUMMARY:
TMS is a non-invasive brain stimulation technique, which can be used to change the activity of a person's brain cells without needles or surgery. In this study, the invesigators are interested in the brain's ability to adapt (also called "neuroplasticity") and regain language functioning after a stroke-specifically, they want to determine whether how a person's brain responds to TMS in the short term can be used to predict how well they will recover language abilities in the long term.

DETAILED DESCRIPTION:
Aphasia is an impairment of language that may occur after a stroke (or other brain injuries). A person with aphasia may experience difficulties speaking, understanding speech, reading, writing, or any combination of these symptoms. Despite advances in understanding of language systems and functional neuroplasticity after brain injury, accurate predictors of aphasia recovery after stroke remain elusive. In order to better understand, predict, and enhance language improvement after stroke, there is a critical need to develop tools that can assess the influence of neuroplasticity on recovery.

Transcranial magnetic stimulation (TMS) is a non-invasive brain stimulation tool that has been used to predict the brain's neuroplastic capacity by assessing physiological responses observed immediately following administration of TMS. Additionally, difference in the physiological response to TMS have been shown to be affected by polymorphism in the gene coding for brain derived neurotrophic factor (BDNF). The current project explores the idea that because neural mechanisms of plasticity are essential determinants of both recovery after brain injury and physiologic response to TMS, magnetic brain stimulation could be employed as an indicator of the capacity for clinically relevant neuroplasticity, and potentially as a predictor of recovery from post-stroke deﬁcits such as aphasia

The goals of this protocol are to 1) explore the utility of theta burst stimulation (TBS), a type of transcranial magnetic stimulation (TMS), as a tool for assessing neuroplasticity in the language system in patients with aphasia due to stroke, 2) and to assess the utility of TBS as a biomarker and predictor of functional recovery in patients with aphasia.

This protocol will encompass two separate but related experiments. In the ﬁrst experiment, the investigators will apply TBS to brain regions that control language functions in aphasic patients in order to determine whether we can induce a transient improvement in naming ability. They will use a statistical model they have developed to categorize patients as either having High Plasticity or Low Plasticity. The investigators will determine whether this distinction predicts which patients are likely to have greater TBS-induced changes in language performance. In the second experiment, in the same patients, the investigators will apply TBS to the motor cortex to elicit changes in motor evoked potentials (MEPs). Using the same model to form matched groups, we predict that MEPs will be more attenuated in High Plasticity groups compared to the Low Plasticity group.

ELIGIBILITY:
Inclusion Criteria:

* Must have Aphasia due to stroke
* Stroke must have occurred at least 6 months ago
* Native English speaker
* Willing & able to have a MRI

Exclusion Criteria:

* Disorders of the brain other than stroke (i.e. tumor, Parkinsons, cancer... etc.)
* History of seizures/ or epilepsy
* Pacemaker or other implanted electronic devices
* Consumption of medications that lower seizure threshold
* History of psychiatric disorders
* History of tinnitus
* Current abuse of drugs or alcohol
* Pregnant or plan to get pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have had one or more strokes and are now experiencing the symptoms of aphasia. Aphasia is a communication disorder which may result in difficulties speaking,understanding speech, or both.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2013-07; Primary Completion 2019-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Transient TBS-induced changes in motor evoked potentials (MEPs) | Up to 2 week
  Single-Pulse TMS will be used to measure MEPs prior to and after stimulation. When measuring MEPs, single pulses of TMS will be administered at approximately 120% of motor threshold, and with a minimum interstimulus interval of 5 seconds. Mean MEP amplitudes will be calculated by averaging the MEP amplitudes generated by 20 pulses. MEP measures will be obtained three times in order to establish a stable baseline. This procedure will be followed by TBS delivered to the optimal site in the motor cortex. TBS will be applied to the region of the primary motor cortex (M1) representing the hand. After TBS, MEPs will be acquired, at 0-, 10-, 20-, 30-, 40-, and 60-min post-stimulation.
Transient TBS-induced changes in language performance | Up to 4 weeks
  Participants will be asked to perform a 40-item picture naming task pre/post TBS stimulation. Stimulation will occur at language cortex and vertex (order will be counterbalanced). Transient changes in naming abilities will be measured directly by assessing naming performance.

SECONDARY OUTCOMES:
Safety and Tolerability of TBS in patient with aphasia | Through study completion
  We will collect the number of patients with TMS-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Roy H Hamilton, MD, MS, Principal Investigator — Neurology
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Lab Website — http://www.med.upenn.edu/lcns/